CLINICAL TRIAL: NCT04695223
Title: Targeting Structural p53 Mutations With Arsenic Trioxide for Intractable Cancer
Brief Title: Arsenic Trioxide for Structural p53 Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Sheng Zang, Department Director, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANTI-P53
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Arsenic Trioxide; p53 Mutations; Refractory Cancer; Intractable Cancer
MeSH Terms: conditions — Neoplasms | interventions — Arsenic Trioxide; Arsenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arsenic Trioxide (Experimental): Arsenic Trioxide (0.16mg/kg,d1-5,ivgtt,28days as a duration) for injection
  Interventions: Drug: Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic Trioxide — Refractory cancer patients without standard-of-care harboring TP53 mutation received Arsenic Trioxide Injection (0.16mg/kg,d1-5,ivgtt,28days as a duration)
  Other Names: As2O3; Arsenic

SUMMARY:
TP53 is the most frequently mutated gene in cancer, but these mutations remain therapeutically non-actionable. Previous study reported arsenic trioxide could rescue structural p53 mutations, endowing p53 mutations with thermostability and transcriptional activity. Under Vivo and Vitro experiments, arsenic trioxide could reactivate mutated p53 to inhibit tumor. This trial aimed to explore the efficacy and safety of arsenic trioxide in refractory cancer patients with structural p53 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Malignant solid tumors diagnosed histologically;
* Solid tumor patients have no any standard choice after multiple line of therapy;
* Next-generation Sequence showed TP53 mutation;
* Expected survival ≥ 1 month;
* ECOG / PS score: 0-2, and the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN); Liver ALT and AST <2.5 × ULN and if liver metastases, ALT and AST <5 × ULN; Serum Cr ≤ 1 × ULN, endogenous creatinine clearance ≥50ml/min
* normal cardiac function
* obtain informed consent

Exclusion Criteria:

* Patient still has standard treatment therapy based on NCCN guidance;
* Patient can not comply with research program requirements or follow-up;
* woman who are pregnant or breastfeeding;
* allergic to any drug in protocol or with contraindications;
* cannot understand or obey the protocol;
* with a history of allergies or intolerability;
* participate in other clinical trials meanwhile;
* any situations that hinder trial existed;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 2 months
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission
Progress Free Survival | Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 2 months
  Time from treatment beginning until disease progression

SECONDARY OUTCOMES:
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 1 months
  Time from treatment beginning until death from any cause
Adverse Effect | Through study completion, an average of 1 months
  Incidence of Treatment-related adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang Y, Song H, Wang Z, Xiao S, Xiang X, Zhan H, Wu L, Wu J, Xing Y, Tan Y, Liang Y, Yan N, Li Y, Li J, Wu J, Zheng D, Jia Y, Chen Z, Li Y, Zhang Q, Zhang J, Zeng H, Tao W, Liu F, Wu Y, Lu M. Repurposing antiparasitic antimonials to noncovalently rescue temperature-sensitive p53 mutations. Cell Rep. 2022 Apr 12;39(2):110622. doi: 10.1016/j.celrep.2022.110622. PMID 35417717